CLINICAL TRIAL: NCT06908590
Title: Heart-to-Heart: A Community Health Worker-Led Intervention to Increase Cardiac Rehabilitation Participation Among Patients With Low Socioeconomic Status
Brief Title: Community Health Worker-Led Intervention to Increase Cardiac Rehabilitation Participation
Acronym: H2H
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00463207; 1K23HL161404 (NIH)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: CVD - Cardiovascular Disease
Keywords: cardiac rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Educational Status; Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H2H Intervention (Experimental): Providing the H2H Intervention to Participants
  Interventions: Behavioral: Education, Providing and Engaging Social Support and Assistance with Health System Navigation

INTERVENTIONS:
Behavioral: Education, Providing and Engaging Social Support and Assistance with Health System Navigation — 1. Introduction to Program and Cardiac Rehab Needs Assessment Education about Cardiac Rehab
  2. Education about CVD and how Cardiac Rehab can help in the participants recovery
  3. Social Support Module
  4. Health System Navigation Module

SUMMARY:
This study is being done to evaluate whether a program called Heart to Heart, that helps patients make a more informed decision about cardiac rehab (CR), is interesting, acceptable to participants, and whether participants would recommend it to others.

DETAILED DESCRIPTION:
This is a prospective, single-institution pilot study to evaluate the acceptability, feasibility and preliminary efficacy of a tailored Community Health Worker (CHW) led intervention to increase CR participation called H2H. Individuals hospitalized with Cardio Vascular Disease (CVD) events (aged 21 and older) will be identified and screened for eligibility from two Johns Hopkins acute care sites into the pilot study. The duration of participation for each participant is up to 6 months from baseline assessments.

All participants will complete a survey at baseline, 3-, and 6-months and will have medical record abstraction conducted performed by the Johns Hopkins (JH) research study team.

For the intervention, participants enrolled in the H2H program will complete between 4 to 8 coaching sessions with the CHW (delivered by telephone and/or video chat) who will provide tailored education, improve or engage the participant's existing social support network, and assistance with health system navigation over a 3-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized with cardiac events and eligible for CR at Johns Hopkins Hospital and Bayview Medical Center. CR eligibility is determined by their treating health care team .
2. Low socioeconomic status defined by Medicaid insurance, or top quartile of the area deprivation index in Baltimore city.
3. Age ≥ 21 years
4. Willing to be audio-recorded

Exclusion Criteria:

1. Formal diagnosis of dementia or cognitive impairment in the Electronic Health Record (EHR) that would prohibit completion of study activities
2. Formal diagnosis of a severe psychiatric disorders by Diagnostic and Statistical Manual (DSM-5) criteria in the EHR that would prohibit completion of study activities (e.g., schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder).
3. Systemic illness limiting longevity (e.g., advanced cancer)
4. Contraindications to CR as assessed by their health care team
5. Unwilling or unable to follow study procedures.
6. Unable to consent
7. Unable to speak or understand English. Assessments including in-depth interviews will be conducted in English.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of H2H intervention as assess by the ability to recruit ≥ 25% of those eligible and the ability to retain ≥ 50% in the study | 3 months
  Proportion enrolled in the H2H among those eligible and approached, and Proportion who complete 4 H2H sessions or enroll in CR
Acceptability as measured by survey of participant satisfaction with H2H | 3 months
  Questionnaire:
  Scores on questionnaire to assess satisfaction. Questions are rated on a Likert scale from 1 (not at all) 5 extremely. There are 6 questions in the rating of the overall program with a total score range 6-30. Acceptability cutoff will be proportion of participants with score ≥ 18. There are 4 questions on the H2H coaching sessions and CHW. The maximum and minimum scores are 4 and 20 respectively. Acceptability cutoff will be proportion of participants with scores ≥ 12.
Acceptability as measured by participant satisfaction (qualitative interview) | 3 months
  A semi-structured interview will be conducted by the research team about the H2H Program overall, and about the coaching sessions with the CHW, to determine the participants' perceptions of the degree to which the intervention was engaging, feasible, acceptable and useful. Recommendations for improving the H2H Program will be solicited. The interviews will take approximately 30-45 minutes. The interviews will be transcribed and analyzed for themes and codes

SECONDARY OUTCOMES:
Change in Cardiac rehab barriers scale | 3 months
  Change in Cardiac Rehab Barriers Scale: 21-item questionnaire that assesses participants perceptions of barriers to CR. Each item is rated on a 5-point Likert Scale, with 1 indicating strong disagreement and 5 indicating strong agreement. This is a validated scale. Score range 21- 105. Higher scores indicate greater barriers to patient enrollment or participation in a CR program.
Change in Patient Activation Measure | 3 months
  13-item questionnaire that assess participant's knowledge, skills, and confidence in managing their own health and healthcare. It is a validated patient related outcome measure. Each item rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Score range is 13-52. Then, this score is transformed to a scale with a theoretical range 0-100, based on calibration tables, with higher Patient activation measure 13 (PAM13) scores indicating higher patient activation
Number of CR sessions attended | 3 and 6 months
  (Preliminary Efficacy) Total number of CR sessions attended. This can range from 0 to 36.

OTHER OUTCOMES:
Number of CHW sessions contacts | 6 months
  (Process Measures of Content Delivery) Number of CHW sessions contacts, where content is delivered, extra contacts, numbers of contacts attempted, number of contacts completed
Duration of CHW sessions contacts (minutes) | 6 months
  (Process Measures of Content Delivery) Duration of coaching session
Number of CHW sessions contacts attempted | 6 months
  (Process Measures of Content Delivery) Number of CHW sessions contacts attempted
Number of CHW sessions contacts completed | 6 months
  (Process Measures of Content Delivery) Number of CHW sessions contacts completed
Change in Health Related Quality of Life as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale | 3 and 6 months
  Change in mean score on the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale
  PROMIS is a 10-item questionnaire that measures a person's global physical and mental health. This is a validated scale.
  Uses a 5-point Likert scale for most items, with a pain intensity item scored on a 0-10 scale (then recoded to a 5-point scale), to assess physical, mental, and social health, producing Global Mental and Physical Health scores.
  The score range for the PROMIS Global Health scales is 0- 100. Higher scores are better.
Change in Depressive Symptoms as assessed by the Patient Health Questionnaire (PHQ)-8 | 3 months
  Change in mean score on the Patient Health Questionnaire (PHQ)-8
  8-item scale that measures depressive symptoms over the past two weeks.
  Each of the eight items on the PHQ-8 is scored on a scale of 0 to 3, with 0 representing "not at all" and 3 representing "nearly every day"
  The total score is calculated by adding up the scores from each of the eight items, resulting in a possible score range of 0 to 24
  A score of 5-9 indicates mild depressive symptoms, 10-14 moderate, 15-19 moderately severe, and 20-24 severe.
Change in Anxiety Symptoms as assessed by the Generalized Anxiety Disorder (GAD7) | 3 months
  Change in mean score on the Generalized Anxiety Disorder (GAD7)
  GAD7 is a 7-item scale those measures anxiety symptoms over the past few days, from not at all to nearly every day.
  Each of the 7 items is scored from 0 to 3, with higher scores indicating greater severity of anxiety symptoms
  A score of 5-9 indicates mild anxiety, 10-14 moderate, 15-19 moderately severe, and 20-21 severe anxiety
  The Generalized Anxiety Disorder-7 (GAD-7) scale has a maximum score range of 0- 21.
Change in Perceived Stress as assessed by the Perceived Stress Scale (PSS10) | 3 months
  Change in mean score on the Perceived Stress Scale (PSS10).
  PSS-10: The PSS-10 is a 10-item questionnaire where each item is scored on a 5-point Likert scale (0 = never, 4 = very often).
  The score range on the Perceived Stress Scale (PSS) is 0-40, with higher scores indicating greater perceived stress.
Change in Physical Activity as assessed by the Telephone Assessment of Physical Activity (TAPA) | 3 and 6 months
  Change in total score on the Telephone Assessment of Physical Activity (TAPA)
  9-item questionnaire that asks the frequency, intensity, and duration of physical activity. This is a validated scale.
  Each question has a 'Yes' or 'No' option. The total score of the first seven items is out of 7; participants choose which question corresponds to their activity level. Any score less than 6 is considered suboptimal. Strength training and flexibility are scored separately (strength training = 1, flexibility = 2, both = 3)
All-cause hospitalization | 6 months
  Hospitalization
All-cause mortality | 6 months
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Lena Matthews, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland